CLINICAL TRIAL: NCT06425120
Title: Effect of Xuesaitong Soft Capsules on Major Risk Factors in Patients With Coronary Heart Disease: a Multicenter, Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Effect of Xuesaitong Soft Capsules on Major Risk Factors in Patients With Coronary Heart Disease
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Jing Li, JingLi, MD, PhD, professor, China National Center for Cardiovascular Diseases
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2023-ZX074
Record Dates: First submitted 2024-05-17; First posted 2024-05-22 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Xuesaitong Soft Capsule (Experimental): Each participant in the Xuesaitong Soft Capsule treatment group will take a daily dose of 1.32g.
  Interventions: Drug: Xuesaitong Soft Capsule
- Placebo (Placebo Comparator): Each participant in the placebo group will take matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Xuesaitong Soft Capsule — Each participant in the xuesaitong soft capsule treatment group will take a daily dose of 1.32g.
  Other Names: LixuwangⓇ
  Arms: Xuesaitong Soft Capsule
Drug: Placebo — Each participant in the placebo group will take matching placebo.
  Arms: Placebo

SUMMARY:
This trials aims to assess, in 240 eligible patients with coronary heart disease, the effects on level of high-sensitivity C-reactive protein (hsCRP) changes from baseline to 12 weeks of Xuesaitong Soft Capsules.

DETAILED DESCRIPTION:
In this multicenter, randomized, double-blind, placebo-controlled trial in patients with coronary heart disease,240 eligible patients aged ≥18 years will be randomized to receive placebo or Xuesaitong Soft Capsules(1.32g/d) and be followed up for 3 months. The primary endpoint of this study is hsCRP change from baseline to 3 months. The secondary endpoint is the changes of following indicators or scores from baseline to 3 months:(Ⅰ)other inflammation indicators except for hsCRP. (Ⅱ) inhibition of platelet aggregation; (Ⅲ)endothelial function indicators; (Ⅳ)blood lipid levels; (Ⅴ) seattle angina questionnaire score; (Ⅵ)36-item short form health survey score. The safety of using Xuesaitong soft capsules in patients with coronary heart disease will also be evaluated. The generalized linear mixed effects model will be used to evaluate the efficacy endpoint for the "full analysis set". For the safety analysis set, Chi-square test will be used to evaluate the safety endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old
2. Chronic coronary artery disease: meet any of the following conditions, and the condition is stable for at least 3 months:

   1. History of myocardial infarction
   2. Have received coronary interventional therapy
   3. There are symptoms of myocardial ischemia (such as chest pain) and objective evidence (stress electrocardiogram or stress myocardial perfusion imaging indicated myocardial ischemia or coronary artery stenosis ≥50% )
3. High-sensitivity C-reactive protein ≥2mg/L
4. Currently taking moderate or above intensity statins lipid-lowering drugs
5. Currently taking antiplatelet drugs
6. Sign informed consent

Exclusion Criteria:

* Patients fulfilling any of the following criteria are not eligible for inclusion in this trial:

  1. Acute coronary syndrome occurred or received percutaneous coronary intervention therapy within the past 3 months
  2. Previously received coronary artery bypass grafting
  3. Stroke occurred within the previous 3 months
  4. Symptomatic heart failure (HF) in the past, or documented left ventricular ejection fraction < 35%
  5. Revascularization or surgical procedures are planned within the next 3 months
  6. Progressive neuromuscular disease, or creatine kinase (CK) levels > 3 times the normal upper limit (ULN)
  7. Lupus, inflammatory bowel disease, severe arthritis and other inflammatory diseases
  8. Immunosuppressants such as cyclosporine, tacrolimus, azathioprine, or systemic steroids are currently being taken or planned during the study
  9. History of hereditary dyslipidemia such as familial hypercholesterolemia
  10. There has been a change in lipid regulation treatment within the past 1 month, or there is a current adjustment plan
  11. History of symptomatic non-traumatic cerebral hemorrhage at any time in the past
  12. History of gastrointestinal bleeding or major surgery within the past 6 months
  13. Use of Xuesaitong soft capsules or preparations containing the main ingredients of Xuesaitong in the past 1 month
  14. There were clear adverse reactions to the main components of Xuesaitong in the past
  15. Active liver disease, or alanine aminotransferase (ALT) levels > 3 times the upper limit of normal (ULN)
  16. Chronic kidney disease, or estimated glomerular filtration rate (eGFR) <60ml/ (min×1.73m2)
  17. Pregnancy or planned pregnancy, or breastfeeding
  18. Malignant tumors, or other serious diseases with an estimated survival of less than 1 year
  19. Mental disorders or communication disorders, cognitive impairment, or other serious medical conditions that may affect study participation
  20. Have participated in or are participating in other clinical trials within the last 1 month
  21. Poor adherence to follow-up or medication is known

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
hsCRP | 12 weeks
  Changes in high-sensitivity C-reactive protein level from baseline at 12 weeks

SECONDARY OUTCOMES:
Other inflammation indicators | 12 weeks
  Changes in levels of interleukin-6, interleukin-10, interleukin-1β, tumor necrosis factor-α from baseline at 12 weeks
IPA | 12 weeks
  Changes in level of inhibition of platelet aggregation from baseline at 12 weeks
Vascular endothelial function | 12 weeks
  Changes in intercellular adhesion molecule-1, von Willebrand factor, and endothelin-1 levels from baseline at 12 weeks
Blood lipid profiles | 12 weeks
  Changes in total cholesterol, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol, small low-density lipoprotein cholesterol, and triglyceride levels from baseline at 12 weeks
Seattle Angina Questionnaire | 12 weeks
  Changes in Seattle angina scores from baseline at 12 weeks
SF-36 | 12 weeks
  Changes in Health Survey Scale (SF-36 Scale) scores from baseline at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jing Li, MD, PhD, Principal Investigator — National Center for Cardiovascular Diseases; Jiamin Liu, MD, Principal Investigator — National Center for Cardiovascular Diseases
Locations (2):
- China (2):
  - Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu

IPD SHARING:
Plan to Share IPD: No